CLINICAL TRIAL: NCT02026037
Title: A Brief Intervention to Reduce PTSD in Acutely Burned Hospital Patients
Brief Title: Reducing PTSD in Hospitalized Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, John Briere, Associate Professor of Psychiatry and Psychology, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CTSI 21-2716-3128
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Stress Disorders; Post-Traumatic; Burns; Brief Psychotherapy; Cognitive Behavior Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Burns | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Brief Treatment for Acutely Burned Patients (BTBP)
  Interventions: Behavioral: Brief Treatment for Acutely Burned Patients (BTBP)

INTERVENTIONS:
Behavioral: Brief Treatment for Acutely Burned Patients (BTBP) — Brief Treatment for Acutely Burned Patients (BTBP) adapts CBT principles that have been validated with non-burn trauma survivors to the treatment of hospitalized burn patients. BTBP consists of three 1 to 1½ hour sessions per week for two weeks, as well as two sessions for family members or partners/spouses.

SUMMARY:
The investigators propose to develop and pilot-test a short-term cognitive-behavioral treatment (CBT) for hospitalized survivors of acute burns, in order to reduce posttraumatic symptoms before they consolidate into long-term posttraumatic stress disorder (PTSD). This is important because approximately one third of burn survivors develop PTSD after discharge. PTSD is associated with extended psychological suffering and a greater need for medical services in the future. Although there are treatments for chronic PTSD, there are far fewer interventions available to treat acute posttraumatic symptoms before they develop into this disorder, and none to date has focused on adult burn survivors. The little research available on other forms of trauma suggests that interventions developed to treat PTSD may be helpful in preventing PTSD when used in the first weeks following a trauma.

The investigators will develop a six-session intervention package for use with patients at the Los Angeles County + University of Southern California Burn Center. The intervention will translate CBT principles that have been validated with trauma survivors, but will be adapted to hospitalized burn patients. After manual development, we will pilot-test this treatment on 15 patients who are medically stable, and not critically ill, intubated, or delirious. Treatment will consist of three 50-minute CBT sessions per week, involving mindfulness-focused relaxation training, graduated exposure to memories of the burn, psychoeducation, and cognitive restructuring. Assessment will include standardized tests of posttraumatic stress, anxiety, and depression, administered at the initiation and termination of treatment, and at one-month follow-up. Also assessed will be number of hospital days to discharge and participant satisfaction with treatment. We will evaluate the overall feasibility of conducting a study on PTSD prevention in burn survivors, as measured by initial recruitment success, subsequent dropout rates at the end of treatment and at the one-month follow-up, and participant satisfaction. These data will then be used to support a subsequent application for funding of a larger-scale randomized clinical trial (RCT) study.

ELIGIBILITY:
Inclusion Criteria:

* Male & female patients at the LAC+USC Medical Center Burn Center
* 18 years of age or older
* English-speaking, able to read & write English
* Expected by the treatment team to require at least 2 weeks of hospitalization
* Willing to participate

Exclusion Criteria:

* Patients who are critically ill; intubated; unable to converse; or delirious
* Cognitively impaired or mentally retarded
* Severely depressed or suicidal
* Psychotic; manic or hypomanic due to a bipolar affective disorder
* Currently demonstrating withdrawal from alcohol or other substances
* Patients whose physical pain level requires medications that would cognitive impair him or her to the point of diminished or impaired functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Posttraumatic Stress-Total (PTS-T) scale of Detailed Assessment of Posttraumatic Stress (DAPS) | 6 weeks

SECONDARY OUTCOMES:
Change from baseline on Beck Depression Inventory | 6 weeks

OTHER OUTCOMES:
Change from baseline on Beck Anxiety Inventory | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Briere, Ph.D., Principal Investigator — University of Southern California; Warren Garner, M.D., Principal Investigator — University of Southern California; Randye J. Semple, Ph.D., Study Director — University of Southern California
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States